CLINICAL TRIAL: NCT05663853
Title: A Multicenter Observational Study for Ex-vivo Evaluation of the Likelihood of Response to an Experimental Tolerance Restoration Therapy in Subjects Diagnosed With Multiple Sclerosis (MS)
Brief Title: An Observational Biomarker Study in Multiple Sclerosis (MS) Patients
Status: Completed | Type: Observational
Sponsor: LAPIX Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LPX641-001
Record Dates: First submitted 2022-12-08; First posted 2022-12-23 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All males and females between 18-70 years of age regardless of their race and ethnicity with a confirmed diagnosis of Primary Progressive Multiple Sclerosis (PPMS), Secondary Progressive Multiple Sclerosis (SPMS), and Relapse Remitting Multiple Sclerosis (RRMS) are invited to participate in this Observational study being conducted across four sites in the US. Since this is an observational study no medication/drug or treatment will be given to the participants. The investigator will be collecting information about the participant's MS disease, its progression, current medications, radiographic scans, and blood samples. This will help the investigator evaluate the biomarkers and new treatment options to better understand the MS disease process.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic disabling disorder of the central nervous system with inflammatory etiology and genetic and environmental factors. It affects females more than males (2-3:1ratio). The National Multiple Sclerosis Society estimates 2.8 million people are affected by Multiple Sclerosis (MS) globally, with around 1 million patients in the US alone.

This is an observational protocol designed to collect clinical and radiographical data and blood samples from patients with a confirmed diagnosis of multiple sclerosis (MS). The blood samples are collected to conduct research on the likelihood of response to LAPIX's novel small molecule therapy and to better understand the MS disease process. Since this is an observational study, no drug or device will be administered to the participants and randomization will not be performed. There will be no alterations/modifications to the current treatment plan or modalities of the enrolled participants. This multicenter study will be conducted across four US sites that will enroll 200 MS patients. The total duration of this observational study (including the screening period and Visit-1) will be 7 days. However, both the screening period and Visit-1 can be combined into a single visit. There will be no follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a confirmed diagnosis of different types of Multiple Sclerosis (MS) namely PPMS, SPMS, and RRMS, by the revised 2017 McDonald criteria.
2. Male or female MS subjects aged 18 -70 years.
3. Body Mass Index (BMI) 18.0-35.0 kg/m2 at screening.
4. Subjects have undergone 1.5T and/or 3T MRI brain and /or spinal cord with or without contrast within the past 6 months.
5. Subject, or their legally authorized representative/guardian, must be willing and able to provide written informed consent prior to initiation of any study procedures.
6. Subjects who are willing and able to adhere to study protocol requirements including but not limited to scheduled visits and laboratory tests.

Exclusion Criteria:

1. Subjects diagnosed with Clinically Isolated syndrome (CIS) which describes the first episode of neurological symptoms that last at least 24 hours caused by inflammation or demyelination in the central nervous system. It usually occurs in young adults and affects optic nerves, the brainstem, or the spinal cord.
2. Subjects with a confirmed diagnosis of NMOSD by the 2015 International Panel for NMO Diagnosis (IPND) criteria.
3. Subjects with a confirmed diagnosis of MOGAD by meeting the following criteria:

   1. Laboratory finding serum positive MOG-IgG by cell-based assay.
   2. Clinical findings of any of the following presentations:

   i)Acute disseminated encephalomyelitis (ADEM) ii)Optic neuritis, including chronic relapsing optic neuropathy (CRION) iii)Transverse myelitis (short or long segment) iv)Brain or brainstem syndrome compatible with demyelination v)Any combination of the above c) Exclusion of the alternative diagnosis.
4. Subjects with Grade-3 lymphocytopenia (<500-200 /mm3 or <0.5-0.2* 10e9/L) over the past 6 months.
5. COVID-19:

   Subject has a known COVID-19 positive status (confirmed by clinical signs and symptoms and/or + ve SARS-CoV-2 NAAT result COVID test) during enrollment.

   OR has had recent COVID-19 vaccination including a booster dose in the past 30 days OR has received anti-viral therapy intended to prevent COVID-19 such as Paxlovid, remdesivir, molnupiravir, interferons, Anti-SARS-CoV-2 monoclonal antibodies, IVIG-SARS-CoV-2, COVID-19 Convalescent plasma, etc. in the past 4-6 weeks.
6. Blood loss of >250 mL or donated blood within 56 days, or donated plasma within 7 days, of study screening.
7. Subjects with acute illness such as fever (body temperature of ≥100.4°F or ≥ 38°C), vomiting, cough, or diarrhea within 48 hours before the screening period. (Upon recovery these subjects can be rescreened / re-enrolled in the study.
8. Recent vaccination with live attenuated vaccines such as influenza, MMR, Herpes zoster, varicella, yellow fever, Rotavirus vaccine, etc., or inactivated vaccines such as Hepatitis A, Rabies vaccine, etc. in the past 30 days.
9. Subject has participated in another investigational study involving any investigational product within 60 days to the start of the study, or within 5 half-lives, of the experimental drug, biologic, or device whichever is longer.
10. Subjects who have been recently diagnosed or have a documented history of HIV or HIV-related disease conditions, hepatitis B or C, or other infectious diseases.
11. History of cancer treatment with either chemo or radiation therapy or both in the past 5 years prior to enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is not based on self-representation of gender identity.
Study Population: Subjects with a confirmed diagnosis of different types of Multiple Sclerosis (MS) namely PPMS, SPMS, and RRMS, by the revised 2017 McDonald criteria.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Collect clinical information pertaining to MS disease | 1 year
  The clinical information includes the date of MS diagnosis, duration of MS, date of last clinical attack, progressive/non-progressive course of the disease, MS medications and treatment modalities, comorbidities, concomitant medications, and vaccination record.
Collect radiographical data | 1 year
  The radiographical data collected but not limited to is the evidence of contrast-enhancing lesions, new T2 lesions, new hyperintense T2 lesions, and hypointense T1 lesions.
Collect patient demographic data | 1 year
  The patient demographic data such as age, sex, race, occupation, and disabilities will be collected.
Evaluate factors affecting the pharmacological response to LAPIX's lead immune-tolerance restoration molecule ex-vivo. | 1 year
  The relationship between ex-vivo exposure to LAPIX's immune-tolerance restoration therapy and pharmacological changes (ex-vivo E-R analysis) will be conducted by the mathematical fitting of the data to an appropriate 3, 4, or 5-parameters E-R model. EC50 and EC90 will be determined by model fitting.
  If potential correlations are found, a more formal statistical analysis may be conducted as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shin, MD,FANA, Principal Investigator — Prof of Neurology MedStar Georgetown University Hospital; Sylvia Klineova, MD,MS, Principal Investigator — Assistant Prof of Neurology Icahn School of Medicine at Mt Sinai; Shiv Saidha, MD,MRCPI, Principal Investigator — Prof of Neurology, Johns Hopkins Hospital, Baltimore MD; Robert Bermel, MD,MBA, Principal Investigator — Director Mellen Center for Multiple Sclerosis, Cleveland Clinic
Locations (4):
- United States (4):
  - The Johns Hopkins University, Baltimore, Maryland
  - MedStar Health, Chevy Chase, Maryland
  - Corinne Goldsmith Dickinson Center for MS, New York, New York
  - Mellen Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No